CLINICAL TRIAL: NCT05297773
Title: Effects of Resistance vs. Aerobic Training on Ki-67 and Other Health-Related Biomarkers: The NEO-Program, a Randomized Controlled Trial on Breast Cancer Patients Undergoing Neoadjuvant Treatment
Brief Title: Resistance vs. Aerobic Training on Breast Cancer Patients Undergoing Neoadjuvant Treatment
Acronym: NEO-Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Collaborators: Faculdade de Motricidade Humana - Universidade de Lisboa (Unknown)
Responsible Party: Principal Investigator, Maria-Joao Cardoso, Head Breast Surgeon - Medical Doctor, Fundacao Champalimaud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Neo-program 2021.02.23; NEO-Program (Other: Fundação Champalimaud)
Record Dates: First submitted 2022-01-25; First posted 2022-03-28 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Exercise; Quality of life; Neoadjuvant treatment; Tumor biology; Physical fitness; Sleep quality
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be followed in a randomized controlled trial conducted during the full duration of neoadjuvant treatment (i.e. 4- to 6-months, depending on patient treatment plan) and two cohorts will be defined: A - breast cancer patients undergoing chemotherapy; B - breast cancer patients undergoing endocrine therapy. Within each cohort, the participants will be divided into three groups: 1) aerobic training; 2): resistance training; 3): control group.
  The intervention is designed to have equal energy expenditure throughout the exercise sessions in both exercise groups (10 kcal/kg/week). All training groups will complete 3 sessions/week. To ensure that both exercise groups are isoenergetic, a portable gas analyzer will be used and blood lactate will be collected.
  Mandatory thematic sessions about several topics such as physical activity guidelines, active lifestyle will be implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Training (Experimental): Three sessions per week during 4-6-months according to each individual treatment plan. Participants allocated in this group will perform moderate-to-vigorous intensity cycling exercise.
  Interventions: Behavioral: Aerobic Training Group
- Resistance training (Experimental): Three sessions per week during 4-6-months according to each individual treatment plan. Participants allocated in this group will perform weight-machine strength exercises of the upper and lower body.
  Interventions: Behavioral: Resistance Training Group
- Control Group (Active Comparator): One session per week of relaxation/stretching.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Aerobic Training Group — The participants will perform continuous cycling at 30%-35% of their heart rate reserve for one month (phase 1: adaptive phase). Then, the intensity will increase every 4-5 weeks (± 5%) up to 80% of heart rate reserve (moderate intensity), depending on the participant's tolerance. An individualized equation establishing the relationship between heart rate, oxygen consumption, and power output will be determined during the cardiorespiratory fitness assessment and used to determine exercise intensity.
  Other Names: AT, moderate continuous cycling
  Arms: Aerobic Training
Behavioral: Resistance Training Group — Initially, and during the first two weeks of the adaptive phase (1-month), the resistance training group will perform one set of 8-12 repetitions (40%-repetition maximum) of 8 exercises for upper and lower body (squat, leg extension, leg curl, deadlift, plank, dead bug, seated row, shoulder press). Then, in the last two weeks, the participants will perform 2 sets of each exercise (45%-repetition maximum). After the adaptive phase, three sets of each exercise will be performed. The initial load will be 50% -repetition maximum increasing up to a maximum of 70%-repetition maximum at the end of the study. Every 4-5 weeks the load will be reviewed and adjusted according to individual.
  Other Names: RT, machine-weight training
  Arms: Resistance training
Other: Control group — The control group will perform a weekly stretching/relaxation session for 45 minutes.
  Other Names: Relaxation/stretching group
  Arms: Control Group

SUMMARY:
A recent consensus study suggested that understanding the impact of exercise on the tumor microenvironment and therapy effectiveness is paramount and should be considered as a research priority. Therefore, the research team intends to address some of the scientific challenges proposed, which represent clear gaps in the current knowledge.

The investigators propose a randomized controlled trial conducted during all neoadjuvant treatment duration that aims to evaluate and compare the effects of two different exercise protocols (aerobic and resistance training) against a relaxation control group on Ki-67% changes as the main outcome in breast cancer patients. Secondary outcomes will be body composition; resting metabolic rate; physical fitness; quality of life, fatigue, depression/anxiety; accelerometry data (physical activity levels, sedentary time); sleep quality; tumor biology (size, hypoxia, and immune profile); glycemic, lipid, and inflammatory profile.

This project will help not only researchers with the design of future exercise intervention protocols but will also help exercise physiologists in the decision-making process when defining training programs. Moreover, the investigators expect that this research program will encourage more cancer patients to exercise. The team expects that patients with breast cancer engaging in structured exercise will show a more marked decrease in Ki-67, tumor size, and hypoxia and increase the tumor-infiltrating lymphocytes (TILs) compared to controls. The investigators anticipate a more noticeable decrease in the preoperative endocrine prognostic index (PEPI) score and in the Residual Breast Cancer (RCB) in both training groups (respectively with hormonal and chemotherapy). Also, frequent declines in physical fitness are expected to be mitigated in exercisers. It is hypothesize that aerobic training will ameliorate cardiorespiratory fitness and fat mass, while the effects of resistance training will be more relevant for muscle strength, muscle mass, and bone health. Both exercise groups will show greater improvements in quality of life, fatigue, depression, anxiety, and sleep quality. Regarding glycemic, lipid, and inflammatory profiles, the investigators expect to see more favorable changes in both training groups, with a more evident decrease in fasting glucose and insulin, HbA1c%, total and LDL-cholesterol, and triglycerides, and the increase in HDL-cholesterol. The increase in C-reactive protein (CRP), tumor necrosis factor -α (TNF-α), interleukin-6 (IL-6), IL-8, IL-1β, IL-1ra, and insulin-like growth factor-1 (IGF-1) and the decrease in brain-derived neutrotophic factor (BDNF), IL-12p70, IL-10, oncostatin M will be smaller in exercise groups.

DETAILED DESCRIPTION:
Exercise plays a crucial role in breast cancer prevention and more recently it appears as a safe, non-pharmacological, and cost-effective adjuvant therapy for cancer. Indeed exercise improves the quality of life, fatigue, physical fitness, and also has a positive impact on tumor intrinsic characteristics.

Most of the studies regarding the effects of exercise in breast cancer patients were performed after surgery or in survivors. Despite being a window of opportunity to study the impact of exercise on biological properties of the tumor, namely on proliferation markers, the investigations conducted during the neoadjuvant period are still scarce and most of the literature derives from animal studies. Although originating from pilot investigations, the initial human-based evidence suggests that exercise interventions are feasible during neoadjuvant therapy and can potentially reduce some proliferation markers such as Ki-67 (i.e. a widely used prognostic marker), induce favorable changes in tumor-related genes, and increase survival.

Power and sample calculations (G-Power, Version 3.1.9.2) are based on an effect size of 0.25 for KI-67 while using ANOVA - repeated measures within-between interactions, a power of 0.80, a significance of 0.05, and an expected dropout of 40%. The calculation yielded a total sample size of 120 participants (60 undergoing chemotherapy and 60 undergoing hormone therapy: 20 participants per group per each treatment). The power and sample calculations were performed using a study that reported the effect of medication on KI-67 since no study has evaluated the effects of an exercise intervention on that variable and has obtained significant results.

Participants will be recruited to take part in an intervention study for breast cancer patients undergoing neoadjuvant treatment. The recruitment will take place at Champalimaud Clinical Center Breast Unit / Champalimaud Foundation.

To improve exercise adherence, the following strategies will be implemented:

* Thematic sessions about several topics such as physical activity (PA) guidelines, active lifestyle, nutrition, the benefits of exercise for breast cancer patients, etc. Each session will last 1-hour (30 minutes presentation + 30 minutes discussion/questions) and will occur once a month. These thematic sessions are mandatory.
* Group activities: once a month, a group activity will be promoted (exercise outdoor sessions, group walk, group dinner, etc.). In these group activities, participants may invite family members to participate.
* The NEO-program website presenting the mission/goals, team members, activities, news and events, contacts, etc.
* Facebook and Instagram account (share information and photos); before the intervention, written consent for image collection will be requested.

The investigator records clinical data, using a paper or electronic case report form (CRF), all data is collected in an online database that is available through the Champalimaud Clinical Center intranet. Participating physicians have a personal account to log in to the registration page and access the electronic CRF. They will have permanent access to their series of patients.

The participating physician ensures the confidentiality, accuracy, completeness, legibility, and timeliness of the data recorded. Data handling and statistical analysis will be done anonymously by the investigator, with the subject identification code list only available to the local investigator (and research nurse if applicable) working in the local center. The code will be based on the birth date and center abbreviation (and not patient initials). The Sponsor will be the owner of the data. Data will be kept for 20 years.

The Participating Investigator and the Participating Site shall treat all information and data relating to the Study disclosed to Participating Site and/or Investigator in this study as confidential and shall not disclose such information to any third parties or use such information for any purpose other than the performance of the Study.

The collection, processing, and disclosure of personal data, such as patient health and medical information are subject to compliance with applicable personal data protection and the processing of personal data legislation (including but not limited to the European Union Directive 95/46/EC).

Champalimaud Foundation takes out the appropriate insurance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically breast cancer (stage 0-III); scheduled for neoadjuvant treatment (cohort A - chemotherapy; cohort B - endocrine therapy)
* Women aged ≥ 18 years; nonpregnant
* Do not be involved in any structured exercise program in the past 6 months
* Medical approval to participate in the study
* Willingness to attend exercise sessions

Exclusion Criteria:

* Treated for any cancer in the past 5 years (except basal cancer)
* Uncontrolled heart disease (heart failure, uncontrolled coronary heart disease, and uncontrolled hypertension, cardiac disease)
* Diabetes mellitus
* Lung condition (chronic obstructive or restrictive pulmonary disease)
* Psychological disorders (dementia, Alzheimer, and Parkinson Disease)
* Severe disability, or other medical condition that prevents from exercise training
* Alcohol or drugs abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Ki67% at the end of the intervention | 4-6 months
  Initial tumor biopsy and the post-neoadjuvant surgical specimen will be evaluated. Pathology evaluation will include the Ki67 assessment.
  The time frame depends on each participant's treatment plan.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) from baseline to T1 and T2 | 4-6 months
  To calculate BMI (kg/m2), Weight and height will be measured on an electronic scale with a stadiometer without shoes wearing minimal clothing to the nearest 0.01 kg/0.1 cm (Seca, Hamburg, Germany). T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes in hip circumferences from baseline to T1 and T2 | 4-6 months
  Hip circumference will be taken around the widest portion of the buttocks. Two measurements (to the nearest 0.1 cm) will be performed and a mean value will be calculated. If the two measurements differ by more than 0.5 cm, a third one will be performed and the two closest measurements will be considered.T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes in waist circumferences from baseline to T1 and T2 | 4-6 months
  Waist circumference will be assessed according to the NIH (horizontal plane at the level of the iliac crest) and World Health Organization (WHO) protocol (midpoint between the lower margin of the last palpable rib and the top of the iliac crest). Two measurements (to the nearest 0.1 cm) will be performed and a mean value will be calculated. If the two measurements differ by more than 0.5 cm, a third one will be performed and the two closest measurements will be considered.T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes in bone mineral density from baseline to T1 and T2 | 4-6 months
  Dual-energy X-ray absorptiometry (GE Lunar Prodigy Primo Hologic, Wisconsin, USA) will be used to estimate bone mineral content/density. T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes in lean body mass from baseline to T1 and T2 | 4-6 months
  Dual-energy X-ray absorptiometry (GE Lunar Prodigy Primo Hologic, Wisconsin, USA) will be used to estimate percentage of lean body mass. T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes in phase angle from baseline to T1, T2, T3, T4, T5, T6 | 4-6 months
  The participants will undergo bioelectrical impedance analysis (BIA) (single frequency, 50 kilohertz (kHz) ± 1%, NutriLAB, Akern) to determine the PhA and body water compartments (total, extracellular, and intracellular). The participants will be measured in a lying position, with legs apart from each other and arms apart from the trunk, so that the medial surface of the limbs will not touch the rest of the body. Four electrodes (2 in each limb) will be placed on the hand and foot of the dominant side, with a distance of 5 cm between both.
  T moments depend on each participant's treatment plan: T1, T2, T3, T4, T5 correspond to 1-, 2-, 3-, 4-, 5-months after the beginning of the intervention, respectively; T6, 6-months (end of the intervention). On those that will undergo a 4-months treatment plan, only T1, T2, T3, and T4 will be performed.
Changes in resting metabolic rate from baseline to the end of the intervention | 4-6 months
  Resting metabolic rate will be measured using indirect calorimetry using a gas analyzer (QUARK resting metabolic rate (RMR) w/ Cardio Pulmonary Exercise Test (CPET), version 9.1, Cosmed, Rome, Italy). The participants will be in a lying position for 30-minutes while using a mask. The first 5-minutes of gas measurement will be discarded. A steady-state period of 5-minutes for oxygen and carbon dioxide volumes (coefficient of variation ≤ 5%) will be used for analyses.
  The time frame depends on each participant's treatment plan.
Changes in peak oxygen content from baseline to the end of the intervention | 4-6 months
  Peak oxygen uptake (VO2 peak) will be determined by an incremental supervised CPET performed on a cycle ergometer. The assessment will start at 20 Watts and then the workloads will increase 10 Watts/min. Cadence: 60-70 rpm. All tests will be monitored using a 12-lead electrocardiogram PC-based acquisition module by a certified cardiologist, and heart rate will be recorded using Omnia software. After the calibration, inspired and expired gases will be continuously analyzed through a gas analyzer (QUARK RMR w/CPET, version 9.1, Cosmed, Rome, Italy). Participants will exercise until at least two of the following test termination criteria are reached: (1) volitional fatigue; (2) respiratory exchange ratio reached 1.1 or higher; (3) predicted maximal heart rate; (4) oxygen uptake do not increase despite increasing workload. Peak oxygen will be determined as the highest 20 seconds average of the last minute.
  The time frame depends on each participant's treatment plan.
Changes from baseline to T1 and T2 in upper limb strength | 4-6 months
  The handgrip strength test (hydraulic calibrated hand dynamometer - JAMAR) as defined by the American Society of Hand Therapists will be performed to assess upper limb strength. 3 isometric repetitions (separated by 1-minute recovery) will be performed in a seated position. The shoulder joint should be adducted and neutrally rotated; the elbow flexed at 90º, and the forearm in midprone neutral position. The mean of the three trials will be calculated. Verbal encouragement will be provided.
  T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes from baseline to T1 and T2 in lower limb strength | 4-6 months
  To evaluate lower limb strength, an isometric mid-thigh pull will be performed while using a force sensor (Chronojump). 3 maximal voluntary repetitions will be performed for 4-5 seconds while receiving a verbal stimulus, with 3 minutes recovery between trials. The bar will be positioned near the thigh and the knees should be positioned at 120º.
  T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Change from baseline to T1 and T2 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Functional Scale Scores | 4-6 months
  The EORTC-QLQ-C30 is a 30-item questionnaire composed of 5 multi-item functional subscales (physical, role, emotional, cognitive , and social functioning), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global quality of life (QOL) subscale, and 6 single item symptom scales assessing other cancer-related symptoms . The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QOL. Responses to all items are then converted to a 0 to 100 scale. For functional and global QOL scales, higher scores represent a better level of functioning/QOL. For symptom-oriented scales, a higher score represents more severe symptoms. T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Change from baseline to T1 and T2 in European Organization for Research and Treatment of Cancer Breast Cancer Module (EORTC QLQ BR23) Functional Scale Scores | 4-6 months
  The EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual functioning, sexual enjoyment, future perspective) and four symptom scales (systemic side effects, breast symptoms, arm symptoms, upset by hair loss). QLQ-BR23 questionnaire employs 4-point scales with responses from 'not at all' to 'very much'. All scores are converted to a 0 to 100 scale. For functional scales, higher scores represent a better level of functioning. T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.

OTHER OUTCOMES:
Changes from baseline to T1 and T2 in Fatigue-FACIT scale | 4-6 months
  Fatigue will be assessed using the 13-item FACIT-fatigue scale for the assessment of fatigue in cancer patients.24 The FACIT-Fatigue is a validated questionnaire that was originally developed for the precise evaluation of fatigue levels in cancer patients with anemia. It consists of 13 questions using a 5 point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). It has been used frequently in the clinical trial setting. Responses to each question are added with equal weight to obtain a total score. The range of possible scores is 0-52, with 0 corresponding to the highest level of fatigue and 52 corresponding to the lowest level of fatigue.
  T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Changes in depression and anxiety from baseline to T1 and T2 | 4-6 months
  Depression and anxiety will be assessed through The Hospital Anxiety and Depression Scale (HADS), which is a 14-item scale composed of two 7-item subscales. Each item could be answered by the patient on a four-point (0-3) response category, which means that each subscale score could range from 0 to 21. Scores below 7 indicate the absence of mood disorder; scores between 8 and 10 suggest a possible mood disorder; scores of 11 or higher indicate problem presence
  T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Subjective Changes in sleep quality from baseline to T1 and T2 | 4-6 months
  Sleep quality will be subjectively assessed through The Pittsburgh Sleep Quality Index. Self-reported usual sleep habits for the majority of days and nights during the past month only. The 19 self-rated and 5 non-self rated questions combined to form seven component scores, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties.
  T1 and T2 depend on each participant's treatment plan: T1, middle of the intervention; T2, end of the intervention.
Objective Changes in sleep quality from baseline to T1 and T2 | 4-6 months
  Sleep quality and efficiency will be objectively and continuously measured by a ballistocardiography through a bed sensor (Emfit Corp., Kuopio, Finland) placed under the mattress at the thoracic level. Sleep score (range 0 to 100) will be determined indicating the quality of sleep. A score higher or around 80 determines a good sleep quality.
  Furthermore, wrist actigraphy will be used.Sleep latency (minutes), sleep efficiency (%), total time in bed (minutes), total time sleeping (minutes), wake before sleep onset (minutes), number of awakenings, and average awakening length (minutes) will be recorded.
Changes from baseline physical activity and sedentary time at T1, T2, T3, T4, T5, T6 | 4-6 months
  Sedentary time and physical activity levels will be assessed by accelerometry (ActiGraph, GT3X model, Fort Walton Beach, FL). All participants will be asked to wear the accelerometer on the right hip, close to the iliac crest. The devices will be activated on the first day (in the morning) and data will be recorded in 60-second epochs. The cut-off values that will be used to define the intensity of physical activity will be as follows: sedentary: < 150 counts·min-1; light: 151-2689 counts·min-1; moderate: 2690-6166 counts·min-1 (corresponding to 3-5.9 Mets); vigorous: ≥ 6867 counts·min-1 (corresponding to ≥ 6 Mets)
  T moments depend on each participant's treatment plan: T1, T2, T3, T4, T5 correspond to 1-, 2-, 3-, 4-, 5-months after the beginning of the intervention, respectively; T6, end of the intervention. On those that will undergo a 4-months treatment plan, only T1, T2, T3, and T4 will be performed.
Changes in tumor size from baseline to the end of the intervention | 4-6 months
  To measure tumor size, radiological techniques (breast magnetic resonance and mammography) will be used. These assessments will be performed at the moment of the diagnosis and before the mammary surgery.
  The time frame depends on each participant's treatment plan.
Changes from baseline tumor hypoxia at the end of the intervention | 4-6 months
  Tumor hypoxia will be assessed using magnetic resonance imaging (MRI) that is already scheduled before and after neoadjuvant therapy. All MRI examinations will be performed on a 3 Tesla clinical scanner equipped with a standard 16-channel breast coil. In addition to a state-of-the-art MRI protocol with T2-weighted, diffusion-weighted (DWI) and dynamic contrast-enhanced (DCE) MR imaging, the following additional sequences will be performed: 1. a multi-echo gradient-echo (GE) sequence for T2*-mapping and a multi-echo spin-echo (SE) sequence for T2-mapping; 2. a dynamic susceptibility contrast (DSC) bolus-tracking perfusion MRI sequence combined with a hybrid single-shot gradient-echo spin-echo (GESE) echo-planar imaging (EPI) readout. These additional sequences will take only more 10 minutes than the standard MRI (30 minutes).
  The time frame depends on each participant's treatment plan.
Changes from baseline tumor infiltrating lymphocytes at the end of the intervention | 4-6 months
  Initial tumor biopsy and the post-neoadjuvant surgical specimen will be evaluated. Tissue microarray blocks, with a sampling of the tumor-infiltrating lymphocytes hotspots from the initial biopsy and surgical specimen material, will be constructed. An immunohistochemical study with CD8+, CD4+, and CD56+ will be performed on the tissue microarray blocks.
  The time frame depends on each participant's treatment plan.
Changes in fasting glucose from baseline to the end of the intervention | 4-6 months
  A certified health care professional will perform all blood sample collections. The participants will be in a seated position and blood samples will be collected from the antecubital vein into dry tubes containing ethylenediaminetetraacetic acid (i.e. anticoagulant). Fasting glucose will be measured.
  The time frame depends on each participant's treatment plan.
Changes in lipid profile from baseline to the end of the intervention | 4-6 months
  A certified health care professional will perform all blood sample collections. The participants will be in a seated position and blood samples will be collected from the antecubital vein into dry tubes containing ethylenediaminetetraacetic acid (i.e. anticoagulant). Lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides) will be measured.
  The time frame depends on each participant's treatment plan.
Changes in inflammatory profile from baseline to the end of the intervention | 4-6 months
  A certified health care professional will perform all blood sample collections. The participants will be in a seated position and blood samples will be collected from the antecubital vein into dry tubes containing ethylenediaminetetraacetic acid (i.e. anticoagulant). Inflammatory marker CRP will be measured. Moreover, the cytokine and immune profile (leptin, adiponectin, BDNF, TNF-α, IL-6, IL-8, IL-10, IL-1ra, IGF-1, oncostatin M) will be assessed using flow cytometry (FACS Calibur, BD Biosciences) with a Cytometric Bead Array technique and ELISA kits.
  The time frame depends on each participant's treatment plan.
Changes in arterial health from baseline to the end of the intervention | 4-6 months
  Arterial function assessment will be performed on the right carotid artery using an ultrasound scanner (MyLab One, Esaote, Genova, Italy) and implemented with a previously validated radiofrequency-based tracking of the arterial wall. Pulse wave velocity will be measure using applanation tonometry using the Complior Analyse software (ALAM Medical, Paris, France).
  The time frame depends on each participant's treatment plan.
Changes in cardiac health from baseline to the end of the intervention | 4-6 months
  Cardiotoxicity will be evaluated through the assessment of resting left ventricular ejection fraction that could be determined using a two- and three-dimensional electrocardiogram. The time frame depends on each participant's treatment plan.
Changes from baseline mitochondrial respiration at the end of the intervention | 4-6 months
  For mitochondrial respiration, the tissue samples will be collected using biopsies at the moment of diagnosis and following the exercise intervention at the moment of surgery (surgical specimen). Mitochondrial respiration assays will be performed using the Oxygraph-2k high-resolution respirometer (Oroboros Instruments, Innsbruck, Austria) at 37º loaded with mitochondrial respiration medium MiR05, and in the range of 200-400 nmol O2/ml.
  The time frame depends on each participant's treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Inês R. Correia, MSc, Study Chair — Faculdade de Motricidade Humana - Universidade de Lisboa
Locations (2):
- Portugal (2):
  - Faculdade de Motricidade Humana - Universidade de Lisboa, Lisbon, Cruz-Quebrada
  - Fundação Champalimaud, Lisbon, Lisbon District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939